CLINICAL TRIAL: NCT00743509
Title: A Phase II Study of Oral Cyclophosphamide and Sirolimus (OCR) in Advanced Sarcoma
Acronym: OCR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2008.049
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Osteosarcoma
Keywords: sarcoma; Cyclophosphamide; Sirolimus; Progressive or recurrent, advanced (unresectable or metastatic) high-grade osteosarcoma, Ewing's or soft tissue sarcoma previously treated with chemotherapy.
MeSH Terms: conditions — Osteosarcoma; Sarcoma; Recurrence; Neoplasm Metastasis | interventions — Cyclophosphamide; Sirolimus

ARMS (1):
- Oral Cyclophosphamide and Sirolimus (OCR) (Experimental): Sarcoma patients were given oral Cyclophosphamide and Sirolimus (OCR) in 28 day cycles.
  Interventions: Drug: Cyclophosphamide and Sirolimus

INTERVENTIONS:
Drug: Cyclophosphamide and Sirolimus — The dose of cyclophosphamide will start at 200 mg (4 tablets) per day on day 1 and will be taken for 7 days every other week of a 28 day cycle.
  Subjects will take 12 mg (12 tablets) of sirolimus on day 1 of treatment as a loading dose followed by 4 mg (4 tablets) daily continuously
  Other Names: Sirolimus (rapamycin, Rapamune)

SUMMARY:
The purpose of this Phase II study will assess the effectiveness of the combination of oral cyclophosphamide and sirolimus in sarcoma patients with relapsed or widespread disease who cannot be cured by surgery, radiation or conventional chemotherapy.

DETAILED DESCRIPTION:
The purpose of this Phase II study you are being asked to participate in will assess the effectiveness of the combination of oral cyclophosphamide and sirolimus in sarcoma patients with relapsed or widespread disease who cannot be cured by surgery, radiation or conventional chemotherapy. Malignant connective tissue tumors of soft tissue and bone (sarcomas) are highly aggressive cancers. There are few available chemotherapy treatments that are active in treating sarcomas. Sarcomas that have metastasized (spread throughout the body) are usually fatal. There is a great need to identify new active drugs to treat metastatic or relapsed sarcomas. Low dose oral daily cyclophosphamide is an established chemotherapy regimen for treatment of malignant and autoimmune disease and is generally well tolerated. Sirolimus is approved for prevention of kidney rejection after transplantation. Temsirolimus, a form of sirolimus, is approved for the treatment of kidney cancer. Sirolimus combined with cyclophosphamide in animal models of sarcoma resulted in significant anti-tumor activity. Tumor and blood samples will be studied to look for known protein targets of the medication to help learn why certain subjects have a favorable response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Progressive or recurrent, advanced (unresectable or metastatic) high-grade osteosarcoma, Ewing's or soft tissue sarcoma previously treated with chemotherapy.
* Bi-dimensionally measurable lesion(s) on cross-sectional radiography, such as computed tomography or magnetic resonance imaging, within 2 weeks of enrollment.
* ECOG/Zubrod performance score 0, 1 or 2.
* Total WBC >3,000, neutrophil count >1,000, platelet count >100,000 within 2 weeks of enrollment.
* Serum creatinine <2.0 times the institutional upper limit of normal (IULN) within 2 weeks of enrollment.
* AST and ALT <2.5 times IULN (or if liver involvement by sarcoma <5 times IULN) within 2 weeks of enrollment.
* Able to ingest oral medications.
* Sexually active women and men of childbearing potential must agree to use an effective method of birth control during the course of the study and for up to 1 month following the last dose of the study drug, in a manner such that risk of pregnancy is minimized. Surgical sterilization, oral contraceptive pills, intrauterine device, double barrier (e.g. condom and diaphragm or spermicidal agents) or abstinence are acceptable forms of birth control.
* Women of childbearing potential must have a negative pregnancy test within 2 weeks prior to treatment.
* Patient must be >16 years of age at the time the consent document is signed by the patient.
* A paraffin block containing sarcoma, either from a previous surgery or recent biopsy, must be available for correlative studies. If a paraffin block containing sarcoma is not available, patients are required to undergo biopsy to obtain tissue for the correlative studies.

Exclusion Criteria:

* Active infection requiring antibiotic treatment.
* Diabetes mellitus not under good control (e.g. hemoglobin A1c > 8% or fasting glucose > 180 mg/dl) with oral agents or insulin.
* Prior treatment with mTOR inhibitor for sarcoma.
* Less than 3 weeks from prior treatment with chemotherapy to start of treatment with cyclophosphamide and sirolimus. Toxicities from prior chemotherapy (except alopecia) should be grade 1 or less before starting treatment with cyclophosphamide and sirolimus.
* Prior radiation less than two weeks since the administration of the last fraction of radiation therapy to the start of treatment. Patients must have recovered from grade 2 or higher radiation-associated toxicities to be eligible. All measurable lesions, which are being targeted, must be outside previously radiated fields or have documented progression at least 6 weeks after completion of radiation.
* Untreated or active CNS involvement by sarcoma.
* Active second malignancy other than carcinoma in situ. Patients with malignancy other than sarcoma in remission are eligible.
* Women who are pregnant or breastfeeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants came in to the University of Michigan Health System outpatient Hematology/Oncology clinic and were consented to participate in this research project after a description of the research was presented by their physician.
  Forty-nine eligible patients were enrolled from September 2008 to December 2009.
Pre-assignment Details: Eligible participants previously treated with chemotherapy underwent screening. Fifty-one patients were consented, 49 enrolled.
Groups:
- Oral Cyclophosphamide and Sirolimus (OCR): Sarcoma patients were given oral Cyclophosphamide and Sirolimus (OCR) in 28 day cycles.
  Cyclophosphamide and Sirolimus : The dose of cyclophosphamide will start at 200 mg (4 tablets) per day on day 1 and will be taken for 7 days every other week of a 28 day cycle.
  Subjects will take 12 mg (12 tablets) of sirolimus on day 1 of treatment as a loading dose followed by 4 mg (4 tablets) daily continuously
Period: Overall Study
Arm/Group | Oral Cyclophosphamide and Sirolimus (OCR)
Started | 49
Completed | 47
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Oral Cyclophosphamide and Sirolimus (OCR)
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants] — Age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 40
    >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 57 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive Without Disease Progression
Description: Patients who were evaluable for response to therapy, alive and without evidence of sarcoma disease progression. Target lesions followed were lesions that had progressed by World Health Organization (WHO) criteria. Disease progression is defined as a greater than or equal to 25% increase in the sum of the product of target lesions, or unequivocal progression of non-target lesions or the appearance of new tumor lesions >10mm.
Time Frame: 6 months
Population: Patients that tolerated and completed at least one 28 day cycle of therapy were considered evaluable
Measure: Number; unit: participants
Arm/Group | Oral Cyclophosphamide and Sirolimus (OCR)
Number analyzed (Participants) | 47
participants | 10

2. Secondary Outcome: Median Overall Survival Time
Description: Median overall duration of survival.
Time Frame: 48 weeks
Population: All patients who completed at least one 28 day cycle
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oral Cyclophosphamide and Sirolimus (OCR)
Number analyzed (Participants) | 47
days | 298 [193 to 408]

ADVERSE EVENTS:
Arm/Group | Oral Cyclophosphamide and Sirolimus (OCR)
Serious Adverse Events (participants affected / at risk) | 17/49
Other Adverse Events (participants affected / at risk) | 36/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cyclophosphamide and Sirolimus (OCR) (N=49)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Death (General disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 1 (1)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Vascular disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Pain (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Other (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cyclophosphamide and Sirolimus (OCR) (N=49)
Hemoglobin (Blood and lymphatic system disorders) | 19 (31)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (17)
Lymphopenia (Blood and lymphatic system disorders) | 25 (42)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (9)
Platelets (Blood and lymphatic system disorders) | 6 (10)
Fatigue (General disorders) | 11 (12)
Fever (General disorders) | 5 (5)
Weight loss (Metabolism and nutrition disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Mucositis/stomatitis (clinical exam) (Investigations) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 4 (4)
Creatinine (Investigations) | 4 (6)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (9)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 3 (4)
Pain (General disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cystitis (Renal and urinary disorders) | 3 (3)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No